CLINICAL TRIAL: NCT05579626
Title: Comparison of Low-Intensity Statin Plus Ezetimibe Versus High-Intensity Statin Therapy on Risk of New-Onset Diabetes Mellitus in Prediabetic Patients With Atherosclerotic Cardiovascular Disease
Brief Title: Comparison of Low-Intensity Statin Plus Ezetimibe Versus High-Intensity Statin Therapy on Risk of New-Onset Diabetes Mellitus (PROVE-DM)
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Seung-Whan Lee, M.D., Ph.D. (Other)
Collaborators: Yuhan Corporation (Industry)
Responsible Party: Sponsor-Investigator, Seung-Whan Lee, M.D., Ph.D., Principal Investigator, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2022-1275
Record Dates: First submitted 2022-10-11; First posted 2022-10-14 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Pre Diabetes; ASCVD
MeSH Terms: conditions — Glucose Intolerance | interventions — Ezetimibe

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high-intensity statin arm (Active Comparator): (high-intensity statin arm): rosuvastatin 20 mg PO qd, once daily
  Interventions: Drug: high-intensity statin arm
- low-intensity statin plus ezetimibe arm (Active Comparator): (low-intensity statin plus ezetimibe arm ): rosuvastatin 5mg /ezetimibe 10mg PO qd), once daily
  Interventions: Drug: low-intensity statin plus ezetimibe

INTERVENTIONS:
Drug: high-intensity statin arm — •high-intensity statin strategy (standard arm): rosuvastatin 20 mg PO qd, once daily
  Arms: high-intensity statin arm
Drug: low-intensity statin plus ezetimibe — •low-intensity statin plus ezetimibe strategy (experimental arm): rosuvastatin 5mg /ezetimibe 10mg PO qd), once daily
  Arms: low-intensity statin plus ezetimibe arm

SUMMARY:
This study is to evaluating the impact of low-intensity statin plus ezetimibe versus high-intensity statin therapy on risk of new-onset diabetes mellitus in patients with atherosclerotic cardiovascular disease who have prediabetes.

DETAILED DESCRIPTION:
Statins [3-hydroxy-3-methylglutaryl coenzyme A reductase (HMG CoA) inhibitors] decreases the risk of death and cardiovascular events in patients with atherosclerotic cardiovascular disease (ASCVD). The cardiovascular benefits of high-intensity compared to low-intensity statin therapy are well demonstrated, and current guidelines recommend high-intensity statin therapy for high-risk patients with ASCVD . However, statin-related side effects are usually dose-dependent, and more frequent in patients receiving high-intensity statin therapy. A meta-analysis of 13 statin trials with 91,140 individuals reported that statin therapy is associated with an increased risk of developing diabetes mellitus (DM) over a 4-year period compared to patients randomized to placebo (odds ratio [OR] 1.09; 95% confidence interval [CI] 1.02-1.17). The high-intensity statin was associated with an increased risk of new onset DM compared with low doses of statins (HR 1.22, 95% CI 1.15 to 1.29). In addition, meta-analysis of five intensive-dose statin trials suggested the likelihood of developing DM is also higher with high-intensity statins compared to moderate-intensity statins in 32,752 subjects over a mean follow-up of 4.9 years (OR 1.12; 95% CI 1.04-1.22).

Prediabetes is a risk factor for ASCVD with a rapidly increasing prevalence worldwide (7.5% in 2019 and projected to reach 8.0% by 2030). Every year about 6.4-12.1% of these people develop diabetes and the risk increase further in the elderly, obese patients, and patients with metabolic syndrome. Considering that the risk of ASCVD increases even before the onset of DM, prediabetes patients need aggressive statin therapy for primary and secondary prevention. However, high-intensity therapy may increase the risk of new-onset DM, especially in patients with pre-diabetes. For this reason, caution is required in determining statin treatment strategies. An effectiveness of statins in reducing cardiovascular events depends on an absolute reduction in low-density lipoprotein (LDL) cholesterol levels and the duration of statin administration A combination therapy of low-dose statin and ezetimibe is an equivalent approach to high-dose statin therapy for decreasing LDL cholesterol level by 50% and achieving LDL cholesterol target level. This strategy is therefore considered attractive to reduce the risk of new-onset DM, and often used because of concerns regarding statin-induced diabetes in pre-diabetic patients. However, there are no data to compare the incidence of new onset DM as a pre-specified primary outcome between two lipid lowering strategies among prediabetic patients with ASCVD. Herein, we designed the study of comparison of low-intensity statin plus ezetimibe versus high-intensity statin therapy on risk of new-onset DM (PROVE-DM), a phase 4 trial involving patients with established atherosclerosis requiring lipid lowering (statin or ezetimibe) agents, comparing a regimen of high-intensity statin (rosuvastatin 20 mg) with the low intensity statin and ezetimibe (rosuvastatin 5 mg plus ezetimibe 10 mg)

ELIGIBILITY:
Inclusion Criteria:

1. Men or women between the ages of 18 and 75 years who have prediabetes

   - Prediabetes consists of impaired fasting glucose (IFG) or impaired glucose tolerance (IGT) or HbA1c
   1. IFG: fasting plasma glucose (FPG) 100 to 125 mg/dL
   2. IGT: 2 hours post-load glucose on the 75g OGTT (oral glucose tolerance test) 140 to 199 mg/dL
   3. HbA1c: 5.7 to 6.4%
2. Patient requiring high-intensity statin due to high risk of a future cardiovascular event if at least one of the following criteria is present via patient history, physical examination, or medical records at the time of screening (Clinically documented ASCVD)

   * acute coronary syndrome (MI or unstable angina)
   * stable angina
   * coronary revascularization (PCI, CABG, and other arterial revascularization procedure)
   * stroke or TIA
   * peripheral arterial disease (<0.9 performed by a vascular lab or angiogram (including CTA) showing ≥ 50%)
   * ThoracoAbdominal Aortic Aneurysm
   * Unequivocally documented ASCVD on imaging

     * significant plaque on coronary angiography on CT (mild, moderate, severe coronary artery disease)
     * significant plaque on carotid ultrasound (mild, moderate, severe carotid disease)
3. Patients who have never taken a statin or who do not have problems adhering to statin therapy
4. Patient must have been on a stable diet prior to randomization and willing to follow the NCEP (national Cholesterol Education Program) TLC (therapeutic lifestyle changes) diet, or equivalent diet, throughout the study.
5. The patient or guardian agrees to the study protocol and the schedule of clinical follow-up, and provides informed, written consent, as approved by the appropriate Institutional Review Board/Ethical Committee of the respective clinical site.

Exclusion Criteria:

1. Patient's pregnant or breast-feeding or child-bearing potential.
2. Concomitant administration of potent inhibitors of CYP3A4 (itraconazole, ketoconazole, protease inhibitors, erythromycin, clarithromycin, telithromycin and nefazodone) or CYP2C9 (relative contraindication not dependent on CYP450 statins).
3. Chronic kidney disease (eGFR<30 ml/min/1.73m2) or dialysis-dependent renal failure
4. Uncontrolled hypothyroidism.
5. Personal or family history of hereditary muscular disorders.
6. History of muscular toxicity with a statin
7. Alcoholism.
8. Hypersensitivity to any of statin and ezetimibe.
9. Hemodynamic unstable conditions at the time of inclusion: cardiogenic shock at the time of randomization, refractory ventricular arrhythmias, or congestive heart failure (New York Heart Association class IV).
10. Any history of hemorrhagic stroke or intracranial hemorrhage within the past 6 months
11. Any surgery requiring discontinuation of statin and/or ezetimibe is planned within 6 months after randomization
12. A diagnosis of cancer (other than superficial squamous or basal cell skin cancer) in the past 3 years or current treatment for the active cancer.
13. Any clinically significant abnormality identified at the screening visit, physical examination, laboratory tests, or electrocardiogram which, in the judgment of the Investigator, would preclude safe completion of the study.
14. Hepatic disease or biliary tract obstruction, or significant hepatic enzyme elevation (ALT or AST > 3 times upper limit of normal) or (Total bilirubin> 2 times upper limit of normal).
15. Life expectancy < 1 years for any non-cardiac or cardiac causes
16. Unwillingness or inability to comply with the procedures described in this protocol.
17. People who have previously been diagnosed with diabetes and are taking lifestyle modification and oral hypoglycemic agent (OHA) or insulin (In woman, gestational diabetes is included)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 2023-03-14 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with New-onset-DM | 36months after randomization
  New onset DM was defined on the the basis of the American Diabetes association guideline if two abnormal test results of following criteria are existed from the same sample or in two separate test samples.
  1. fasting plasma glucose (FPG) ≥126 mg/dL (7.0 mmol/L). Fasting is defined as no caloric intake for at least 8 hours OR
  2. 2 hour plasma glucose during a 75 g oral glucose tolerance test (OGTT) ≥200 mg/dL (11.1 mmol/L) during OGTT. The test should be performed as described by the WHO, using a glucose load containing the equivalent of 75-g anhydrous glucose dissolved in water OR
  3. HbA1C ≥6.5% (48 mmol/mol). The test should be performed in a laboratory using a method that is NGSP (National Glycohemoglobin Standardization Program) certified and standardized to the DCCT (Diabetes Control and Complication Trial) assay.
Number of Participants with death | 36months after randomization
  Major adverse cardiac events are defined as all-cause death

SECONDARY OUTCOMES:
Composite cardiovascular safety | 36months after randomization
  death from cardiovascular cause, non fatal myocardial infarction of nom fatal stroke
Any arterial revascularization | 36months after randomization
  Any arterial revascularization (carotid, coronary aorta or peripheral artery) Any arterial revascularization (carotid, coronary aorta or peripheral artery)
Any potential side effect | 36months after randomization
  Any potential side effect
Each component of the diabetes-mellitus diagnosis criteria | 36months after randomization
  Each component of the diabetes-mellitus diagnosis criteria
All cause mortality | 36months after randomization
  All cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Whan Lee, MD, Principal Investigator — Asan Medical Center
Locations (31):
- South Korea (31):
  - Bycheon Sejong Hospital, Bucheon-si
  - Gyeongsang National University Changwon Hospital, Changwon
  - Chungbuk National University Hospital, Cheonju
  - Gangwon National University Hospital, Chuncheon
  - Daegu Catholic University Medical Center, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - Yungnam universury Hospital, Daegu
  - Chungnam National University Sejong Hospital, Daejeon
  - Konyang University Hospital, Daejeon
  - the Catholic University of Korea, Daejeon St. Mary'S Hospital, Daejeon
  - Gangneung Asan Hospital, Gangneung
  - Chonnam National University Hospital, Gwangju
  - Inje University Haeundae Paik Hospital, Haeundae
  - Hallym University Dongtan Sacred Heart Hospital, Hwaseong-si
  - Gachon University Gil Medical Center, Incheon
  - Jeju National University Hospital, Jeju City
  - Gyeongsang National University Hospital, Jinju
  - Chungnam National University Hospital, Jungnam
  - Dong-A Medical Center, Pusan
  - Inje University Busan Paik Hospital, Pusan
  - Kosin University Gospel Hospital, Pusan
  - Pusan National University Yangsan Hospital, Pusan
  - Asan Medical Center, Seoul
  - Catholic University of Korea, Seoul ST. Mary's Hospital., Seoul
  - Ewha womans university seoul hospital, Seoul
  - Kangdong Sacred Heart Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - The Catholic Univ. of Korea Eunpyeong St. Mary's hospital, Seoul
  - VHS Medical Center, Seoul
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon
  - Ulsan university hospital, Ulsan

IPD SHARING:
Plan to Share IPD: No